CLINICAL TRIAL: NCT03669978
Title: Endovascular Procedures With Computer Assistance in the Chronic Occlusive Arthritis of the Lower Limbs on the Femoro-popliteal Stage.
Acronym: PANORAMIC
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3070
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Occlusive arthritis; bone panorama; arterial panorama
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic occlusive arthritis of the Lower Limbs: Patients with chronic occlusive arthritis of the Lower Limbs with lesions on the femoro-popliteal stage and candidates for endovascular treatment of these lesions.
  Creation of a bone and arterial panorama using EndoNaut® software.
  Interventions: Procedure: Creation of a bone and arterial panorama using EndoNaut® software.

INTERVENTIONS:
Procedure: Creation of a bone and arterial panorama using EndoNaut® software. — The routine care procedure begins with staged injections of contrast medium to provide a map of the lesions. The lesions are then treated by angioplasty with or without stenting.
  New injections of contrast product are made to control the results of the treatment.
  As part of this pilot study, the assistive software and its interface will be linked and with the mobile C-arm X-ray system. Scopic images and angiograms will be retransmitted to be processed by the EndoNaut® software.
  Other Names: EndoNaut® software.

SUMMARY:
Pilot study to assess the feasibility of creation of a bone and arterial panorama by 2D-2D registration technique during endovascular femoro-popliteal procedures with a mobile C-arm X-ray system using EndoNaut® software.

DETAILED DESCRIPTION:
The aim of this study is to show that it is possible to give a complete image of the area to be operated by the surgeon by creating a complete bone and arterial panorama of the femoro-popliteal axis with 2D-2D registration techniques. This study should have a clinical impact for the patient and caregiver. With this technique, we expect a reduction in the irradiation of the patient and the caregivers, a decrease in the volume of injected contrast product and a decrease in operating time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial disease of the lower limbs, all clinical stages, lesions of the femoro-popliteal stage and candidates for endovascular treatment of these lesions.
* Major patients
* Patients not opposed to their participation in the study

Exclusion Criteria:

* Patients requiring conventional surgical revascularization.
* Patient under legal protection (guardianship, safeguard of justice).
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic occlusive arthritis of the Lower Limbs with lesions on the femoro-popliteal stage and candidates for endovascular treatment of these lesions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Quantification of the registration errors | At the inclusion day
  The 2D-2D registration is driven by an error index (intrinsic software criterion) given by the software at the end of the registration process
Volume of contrast product used during the routine care procedure (ml) | At the inclusion day
  Volume are reported in mL
Irradiation parameters: evaluation of the Fluoroscopy duration (min) | At the inclusion day
  Parameter given by the X-ray imaging device
Irradiation parameters: dose-area quantification (mGy/m2) | At inclusion
  Parameter given by the X-ray imaging device
Irradiation parameters: measurement of air Kerma (mGy) | At the inclusion day
  Parameter given by the X-ray imaging device
Irradiation parameters: evaluation of the number of required angiograms | At the inclusion day
  Parameter given by the X-ray imaging device
Operating time (min) | At the inclusion day
  Delay between the beginning (patient anesthesia) and the end (patient transferred to post interventional care room) of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Kaladji, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes Univesity Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No